CLINICAL TRIAL: NCT06107153
Title: Effect of Short-term Basal Insulin Initiation in Newly Diagnosed Type 2 Diabetes on 1-year Glycemic Control
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Basrah (Other)
Responsible Party: Principal Investigator, Haider Ayad Alidrisi, Assistant professor, University of Basrah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Insulin in type 2 diabetes
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Type2diabetes
MeSH Terms: interventions — Insulin Glargine; saxagliptin; Pioglitazone

STUDY DESIGN:
Intervention Model Description: Inclusion criteria:
  1. New diagnosed T2DM with an age of 18 years and above.
  2. HbA1c of equal to or more than 9% and or random serum glucose equal to or more than 300 mg/dl.
  The study will compare the effect of two strategies for glucose control over one year. First, two-week basal insulin and combination glucose-lowering drugs. Second, combination glucose-lowering drugs
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- basal insulin plus glucose lowering drugs (Active Comparator): New diagnosed T2DM with an age of 18 years and above. HbA1c of equal to or more than 9% and or random serum glucose equal to or more than 300 mg/dl.
  Agree to start basal insulin for two weeks
  Interventions: Drug: Insulin Glargine 100 UNT/ML Pen Injector [Lantus]; Drug: Saxagliptin 2.5 mg/ Metformin Hydrochloride extended release 1000 mg; Drug: Pioglitazone 30mg
- glucose lowering drugs only (Active Comparator): New diagnosed T2DM with an age of 18 years and above. HbA1c of equal to or more than 9% and or random serum glucose equal to or more than 300 mg/dl.
  Refuse to start basal insulin.
  Interventions: Drug: Saxagliptin 2.5 mg/ Metformin Hydrochloride extended release 1000 mg; Drug: Pioglitazone 30mg

INTERVENTIONS:
Drug: Insulin Glargine 100 UNT/ML Pen Injector [Lantus] — Insulin is given as glargine U100 at bedtime in a dose of 10 units. The patients will be given instruction to up-titrate the insulin by adding two units every two days with an aim to reach fasting blood glucose (FBG) between 80 - 130 mg/dl using a home glucometer. And to down-titrate the insulin by subtracting two units when the FBG is below 80 mg/dl. The patients continued on basal insulin for two weeks or less when FBG is persistently below 100 mg/dl on a dose of 10 units of insulin Glargine.
  Other Names: Lantus
  Arms: basal insulin plus glucose lowering drugs
Drug: Saxagliptin 2.5 mg/ Metformin Hydrochloride extended release 1000 mg — Saxagliptin 2.5 mg/ Metformin Hydrochloride extended release 1000 mg
  Other Names: Kombiglyze
Drug: Pioglitazone 30mg — Pioglitazone 30mg
  Other Names: Actos

SUMMARY:
In this study, we aim to explore the beneficial effect of early short-term (two weeks), self-titrated, basal-only insulin therapy on the degree of glycemic control over 1-year follow through a prospective cohort.

DETAILED DESCRIPTION:
Despite the development of new drugs and therapeutic strategies for treating type 2 diabetes mellitus (T2DM), achieving long-term glycemic control remains a challenge. Results from the United Kingdom Prospective Diabetes Study (UKPDS) suggest that deterioration of glycemic control can be largely attributed to progressive β-cell loss, irrespective of the nature of pharmacological intervention. Therefore, treatments that can preserve or improve β-cell function are of great interest in the field of T2DM therapeutics. Some studies have shown that short-term intensive insulin therapy in patients newly diagnosed with T2DM produces beneficial effects on β-cell function, glycemic control, and rate of remission within 1 year. However, these studies applied complex regimes for insulin initiations that require frequent follow-up and are difficult to accept as initial therapy for T2DM.

ELIGIBILITY:
Inclusion Criteria: (must have)

* Newly diagnosed type 2 diabetes mellitus on no glucose-lowering drugs and
* Either hemoglobin A1c equal to or more than 9% and/or random blood glucose equal to or more than 300 mg/dl.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus,
* Urine ketone dipstick + and above at baseline or anytime throughout the study.
* Pregnancy.
* Current or recent steroid use.
* History of coronary heart disease and heart failure.
* GFR less than 60 mL/min/1.73 m2.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c less than 7% | three months
  Percentage of patients with hemoglobin A1c of less than 7%
Hemoglobin A1c less than 7% | six months
  Percentage of patients with hemoglobin A1c of less than 7%
Hemoglobin A1c less than 7% | twelve months
  Percentage of patients with hemoglobin A1c of less than 7%
Change in hemoglobin A1c | three months
  mean change in hemoglobin A1c
Change in hemoglobin A1c | six months
  mean change in hemoglobin A1c
Change in hemoglobin A1c | twelve months
  mean change in hemoglobin A1c

SECONDARY OUTCOMES:
Hypoglycemia | two weeks
  Prevalence of capillary blood glucose less than 70 mg/dl by serial monitoring using home glucometer.

CONTACTS AND LOCATIONS:
Overall Officials: Haider A Alidrisi, MD, Principal Investigator — Faiha Specialized Diabetes, Endocrine, and Metabolism Center, University of Basrah, College of Medicine
Locations (1):
- Faiha Specialized Diabetes, Endocrine, and Metabolism Center, Basra, Iraq

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Weng J, Li Y, Xu W, Shi L, Zhang Q, Zhu D, Hu Y, Zhou Z, Yan X, Tian H, Ran X, Luo Z, Xian J, Yan L, Li F, Zeng L, Chen Y, Yang L, Yan S, Liu J, Li M, Fu Z, Cheng H. Effect of intensive insulin therapy on beta-cell function and glycaemic control in patients with newly diagnosed type 2 diabetes: a multicentre randomised parallel-group trial. Lancet. 2008 May 24;371(9626):1753-60. doi: 10.1016/S0140-6736(08)60762-X. PMID 18502299
- [Background] Ilkova H, Glaser B, Tunckale A, Bagriacik N, Cerasi E. Induction of long-term glycemic control in newly diagnosed type 2 diabetic patients by transient intensive insulin treatment. Diabetes Care. 1997 Sep;20(9):1353-6. doi: 10.2337/diacare.20.9.1353. PMID 9283777
- [Background] Li Y, Xu W, Liao Z, Yao B, Chen X, Huang Z, Hu G, Weng J. Induction of long-term glycemic control in newly diagnosed type 2 diabetic patients is associated with improvement of beta-cell function. Diabetes Care. 2004 Nov;27(11):2597-602. doi: 10.2337/diacare.27.11.2597. PMID 15504992
- [Background] Ryan EA, Imes S, Wallace C. Short-term intensive insulin therapy in newly diagnosed type 2 diabetes. Diabetes Care. 2004 May;27(5):1028-32. doi: 10.2337/diacare.27.5.1028. PMID 15111515